CLINICAL TRIAL: NCT01507025
Title: The Effect of Hinge Location on Corneal Sensation and Dry Eye After LASIK: A Systematic Review and Meta-analysis
Status: Completed | Type: Observational
Sponsor: Yifan Feng (Other)
Collaborators: Wenzhou Medical University (Other)
Responsible Party: Sponsor-Investigator, Yifan Feng, Study Director, Wenzhou Medical University
Organization: Wenzhou Medical University (Other)
Other Study IDs: Y20110045
Record Dates: First submitted 2012-01-05; First posted 2012-01-10 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Dry Eye
Keywords: hinge position; dry eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- horizontal flap: patients were scheduled to undergo LASIK and with horizontal flaps(nasal- or temporal-hinge)
- vertical flap: patients were scheduled to undergo LASIK and with vertical flaps(superior- hinge)

SUMMARY:
The purpose of this study is to investigate the possible effect of hinge location on corneal sensation and dry eye syndrome after laser in situ keratomileusis (LASIK).

DETAILED DESCRIPTION:
Dry eye symptoms are a frequent postoperative complication of laser in situ keratomileusis (LASIK). Although estimates of the incidence of dry eye syndrome vary widely, from 3% to 59%, almost all patients will have transient dry eye during the immediate postoperative period.Because of the variability in corneal innervation patterns, altering flap characteristics in LASIK may affect postoperative corneal sensation and dry-eye disease. Some studies have reported that postoperative corneal sensation may be higher and recovery faster in eyes with horizontal flaps (nasal- or temporal-hinge) than in eyes with vertical flaps (superior- hinge). However, some other studies have not established an association between corneal sensation and hinge position. This study reviewed the published literature and performed a meta-analysis aimed to investigate the effects of hinge location on corneal sensation and dry-eye symptoms after LASIK.

ELIGIBILITY:
Inclusion Criteria:

1. each trial should be a prospective randomized controlled clinical trial (RCT),
2. the age of patient population should be over 18 years

Exclusion Criteria:

1. non-randomized controlled trials
2. patients who had had a previous ophthalmic surgery or ocular surface disorders
3. the raw data was not completed

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients were scheduled to undergo LASIK and randomized to different hinge locations
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2011-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Corneal sensitivity | 6 months
  Change of corneal sensitivity by using the Cochet-Bonnet esthesiometer,we chose to analyze results at 1 week and 1-, 3-, 6-month postoperatively.
Tear break-up time | 6 months
  Change of tear break-up time at 1 week and 1-, 3-, 6-month postoperatively
Schirmer's I test | 6 months
  Change of Schirmer's I score at 1 week and 1-, 3-, 6-month postoperatively

SECONDARY OUTCOMES:
Corneal fluorescein staining | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yifan Feng, MD, Principal Investigator — Eye Hospital, Wenzhou Medical College, China
Locations (1):
- Wenzhou Medical College, Wenzhou, Zhejiang, China

REFERENCES:
- [Derived] Feng YF, Yu JG, Wang DD, Li JH, Huang JH, Shi JL, Ye T, Wang QM, Zhao YE. The effect of hinge location on corneal sensation and dry eye after LASIK: a systematic review and meta-analysis. Graefes Arch Clin Exp Ophthalmol. 2013 Jan;251(1):357-66. doi: 10.1007/s00417-012-2078-5. Epub 2012 Jun 15. PMID 22752222